CLINICAL TRIAL: NCT07145632
Title: APP-based Medical Device for Education and Training of Inhalation Technique
Acronym: APPETITE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Björn Nordlund, Senior Lecturer, Associate Professor, RN, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CIV-ID: 23-06-043273
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Asthma (Part 1); COPD
Keywords: Management; Inhaler technique; Metered Dose Inhaler - MDI; Dry Powder Inhaler - DPI
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Two-armed, parallel-designed, individual single-blinded stratified randomised controlled trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Each of the 80 subjects is stratified to block of 4 numbers according daily used inhaler of (1) DPI, (2) MDI or (3) both MDI/DPI. Simple randomisation (1 to 1) will be applied in each block and at each study site. The randomisation will be blinded for the evaluator at 6-12 week visit, which practically means that not the same study personnel will do the baseline randomisation and the final 6-12 weeks assessment of inhalation technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (No Intervention): The comparator is standard assessment and instructions of inhalation technique while healthcare personnel review patient using their inhaler (DPI or MDI) or similar training device without medication.
- Intervention (Experimental): The potential clinical benefit of using an app-based approach for education and training of inhalation technique is to make the support more accessible for patients to use at home or whenever patients feel inhalation support is needed. Another potential benefit and novelty are the objective assessment of inhalation techniques regarding PIF, time to PIF and inspiration time, which is not possible to precisely assess in standard assessment of inhalation technique.
  Interventions: Device: App-based education and training of inhalation technique

INTERVENTIONS:
Device: App-based education and training of inhalation technique — The use of MDI or DPI requires different inhalation techniques and flows, which makes correct inhalation technique more challenging if patient use different types of inhaler devices. Healthcare providers may assess inhalation technique by observation and in addition PIF may be measured by manual meter. However, this does not capture all relevant information about patient's ability to correctly inhale medication and handle prescribed inhaler(s) and do not give instant and automated feedback on the inhalation technique to user. For instance, DPI users should reached a sufficiently high PIF within the first 0.4 seconds [18] and MDI users inhalation time should exceed 4 seconds in adults (2-3 seconds in children) in order to optimize lung deposition of the aerosol during a low PIF [19]. The app-based inhalation medical device gives automated feedback on inspiratory flows that are specific DPI and MDI devices.
  Arms: Intervention

SUMMARY:
Primary aim: To investigate if app-based education and training of inhalation technique improves the rate of successful inhalation techniques compared with control group at 6-12 weeks follow-up visit.

Secondary aims: To evaluate the feasibility, usability, and safety of the investigational during the study period.

Study design: Two-armed, parallel-designed, individual single-blinded stratified randomisation by inhaler (DPI/MDI/both DPI and MDI) controlled trial with assignment (1:1) to (1) standard care and app-based education and training of inhalation technique or (2) standard education of inhalation technique over 6-12 weeks.

Subjects: Subjects from the age of 16 years with documented diagnosis of asthma and/or COPD, daily treated with dry powder inhaler (DPI) or metered dose inhaler (MDI), or both, will be invited to voluntarily participate. Exclusion criteria is age <16 years, no access to use BankID or similar electronic personal identification service, not using smartphone of type Android or iPhone, plan to stop use DPI and/or MDI the following 6-12 weeks from inclusion. No able to independently handle and inhale through DPI or MDI device.

Total sample size: Eighty subjects (females and males) with daily treatment for COPD or asthma will be sufficient, based on the assumption of 25% percentage improvement in success rate of correct inhalation technique in the interventional group compared with control group (75% versus 50%) with 80% power at 5% significance level, including dropouts at 6-12 weeks follow-up visit.

Intervention: At the baseline visit patients will be randomised to app-based intervention consisting of education and training of inhalation technique of all inhalers used on daily basis (the inhalation app-module). Stratified randomisation based on type of inhaler(s); MDI, DPI or both MDI and DPI will be applied. The intervention is the inhalation app-module, which is a medical device that is embedded the AsthmaTuner app. The AsthmaTuner app is a CE-marked cloud-based system, provided by MediTuner AB in Stockholm, Sweden. The intervention group will be instructed to use the inhalation app-module on daily basis to improve their inhalation technique.

Control group: Standard education of inhalation technique using list of standardised criteria and non-app-based education of inhaler technique.

Endpoints: Primary endpoint is the rate of subjects with successful inhalation techniques based on subjective critical endpoints (CIP Table 2) and the following objective endpoints at the 6-12 weeks follow up visit:

* DPI: PIF > 30 L/Min, time to PIF <0.5 seconds measured with the investigational device.
* MDI: inspiration time (> 3 seconds) and PIF less than 60 L/Min measured with the investigational device.

Procedures: At baseline, a trained respiratory nurse will subjectively assess and train each patient's inhalation technique according to defined criteria of device handling (standard education). The AsthmaTuner app is downloaded to a smartphone or tablet computer (Ipad) that is wirelessly (Bluetooth) connected to a home spirometer. In this study the Bluetooth spirometer AsthmaTuner from MIR will be used. Education and training of inhalation technique will include measurement of inhalation flow with an adjustable resistance mounted on the spirometer, Airflow Trainer (MIR). The app gives instruction to set the resistance, so it corresponds to the selected inhaler. Questionnaires and interviews will collect information about the feasibility, safety and experienced usability of the investigational device.

Analysis: The rate of subjects with successful inhalation technique at 6-12-week visit determined by fulfilling objective and subjective critical endpoints in intention-to-treat approach. The effect of using the inhalation app-module will be analysed with logistic regression analysis across randomisation groups. The secondary analysis of feasibility and the experienced benefit of using the inhalation app-module in clinical practice and for patient's education and training of inhalation technique is estimated on a Likert scale from 1 (not at all) to 5 (strongly agree) and presented as mean and median scores.

DETAILED DESCRIPTION:
Introduction:

Worldwide COPD and asthma are prevalent diseases causing death, health problems, impaired quality of life and high costs for individuals and society. Pharmacological therapies for respiratory diseases are commonly delivered by inhalers allowing for lung deposition of the medication. Guidelines for chronic obstructive pulmonary diseases (COPD) and asthma address that patients should receive regular education and correction of inhalation technique. Acceptable inhalation technique is an effective prevention of uncontrolled symptoms and exacerbations for both asthma and COPD. Therefore, education of inhalation technique is a prerequisite to ensure good treatment response. The education of inhalation technique is usually given by nurses, pharmacists or medical doctors and includes training and demonstration of inhaler use and correction of errors at clinical appointment, by observing if patient correctly can manage critical steps of getting the inhaler ready for inhalation by shaking the inhaler, remove the cap, execute the dose correctly and hold breath after inhalation.

Different inhaler devices have different properties with regards to inspiratory resistance and flow to ensure drug deposition in the lungs. Patient's ability to breath in and the internal resistance of the inhaler affects if drug particles will reach the inflammatory of lungs. Particularly, children, and patients with reduced lung function, e.g. during acute exacerbation, risk not being able to inhale properly. Furthermore elderly, irrespectively of COPD could also have compromised ability to generate a sufficient inspiratory flow. Therefore, when prescribing a new inhaler for treatment it is important to evaluate the most appropriate inhaler device for the patient. Overall, there are two major groups of inhalers, dry powder inhaler (DPI) or metered dose inhaler (MDI), with different properties regarding inhalation technique. MDI requires the patient to breath in the drug slowly, and DPI require a more forceful inhalation. A critical challenge is therefore to assess if the inspiratory flow agrees with specific requirement of particular inhaler in use. Although different types of DPI exist (eg. Turbuhaler, Diskus, Novolizer, Breezhaler), generally an airflow is generated through the DPI during inhalation if the breath in flow is sufficiently strong the medication powder leaves the inhaler and enters the mouth and airway. When inhaling, the resistance of the DPI generates a pressure drop and the drug particle are released. The inspiratory outcomes determining optimized lung deposition are the peak inspiratory flow (PIF), the inhalation time, as well as the time to PIF. Late PIF and low volume increases the risk that limited amount of drug particles reaches the lungs, instead, are deposited in the mouth, which can explain poor treatment response.

In view of available literature, clinicians are confronted to control that patient handle their inhalator and generate sufficient high inspiratory flow rate for optimal lung deposition before prescribing DPIs. Inspiratory flow rate can be assessed with the mechanical devices. This is a hand-held manual meter that enables assessment of PIF through adjustable resistance selected for a relevant inhalator (DPI or MDI). Additionally, app-based digital devices could provide even more extensive and detailed characterisation of patient's ability to perform acceptable inspiratory flows regarding pre-specified outcomes of PIF, time to PIF, and flow over time, to ensure optimal lung deposition of the inhaled drug and for evaluation of treatment response. App-based digital device may offer patient's a simpler support for education and training of inhalation technique. Therefore, we have developed an app-based medical device for improving inhalation techniques. The concept of the device consists of app-based materials for education and a CE-marked wireless spirometer (in this study, MIR AsthmaTuner) and CE-marked Airflow Trainer (MIR) to simulate the internal resistance of the common inhalers in use (DPI or MDI). To determine if patient can fulfil acceptable inspiratory flows of millilitres (mL) per second (s), PIF (flow/min), time to PIF (s), inhalation time (s), but others such as area under the curve, and inhalation flow acceleration may be added in the future.

The investigational device is a separate module, inhalation app-module, embedded in the Cloud-based CE-marked system called AsthmaTuner. Our hypothesis is that provided education and training with the medical device measurement will improve the patients' ability to correctly use their inhalers over time. Thus, the aim of this study is to assess the effect of app-based medical device for education and training on inhalation techniques at 6-12 weeks follow-up visit in subjects with asthma and COPD. Secondary aim is to evaluate if the medical device is feasible to use in clinical practice. The study endpoints are peak inspiratory flow (PIF), time to PIF, flow (litre per min), inhalation time (seconds) and breath hold (seconds) divided by DPI and MDI, together with assessment of how the patient handles their inhaler according to a set of critical criteria. Patients treated for COPD or asthma in primary or secondary care will be invited to participate in a two-armed stratified randomised controlled blinded study (RCT) over 6-12 weeks.

The patient will download AsthmaTuner to their smartphone that connects to a Bluetooth spirometer (in this study, MIR AsthmaTuner). Inhalation test through Airflow Trainer, an adjustable resistance mounted on the home spirometer (Airflow Trainer), determines if the inhalation flow agrees with the endpoints for the inhaler used by study subject. The expected results of this trial will allow us to determine if app-based inhalation device improves inhalation technique compared with standard care. The goal of this project is to provide sufficient information for a CE-marked product of the inhalation app-module. The study will be performed by Karolinska Institutet (KI), B. Nordlund research group, also being the sponsor, but supported technically and intellectual expertise from Astra Zeneca and MediTuner AB (the owner of AsthmaTuner).

Description of the investigational device:

The investigational device is the inhalation app-module which will be investigated in this clinical study, version number later than 5.4.13.5. In this study, it will be used in combination with the MIR AsthmaTuner spirometer and Airflow Trainer (adjustable resistance). The inhalation module starts with patients selecting their inhaler type (DPI or MDI). This leads to written instructions which show patients how they should inhale their medication. The patient is then forwarded to the training part of the module, which allows a patient to inhale through their spirometer which is fitted with the Airflow Trainer (MIR). The patient will be able to see how their inhalation went and will pass or fail the training. A potential benefit of the app-based investigational device is the education patients receive about the medication they take. Patients cannot reach the status of 'medication mastered' until they have also completed two quizzes. The first quiz teaches foundations of asthma or COPD (or both if patient has both diagnoses) while the second quiz touches on more advanced topics within the diseases and tips for effectively managing them daily. The inhalation flow is measured by the wireless spirometer (MIR AsthmaTuner), using connecter (Airflow Trainer) for creating inspiratory flow resistance that corresponds to resistance of the prescribed inhalator as presented in Appendix 2.

The product description and regulatory classification of AsthmaTuner according to MDR is class 2b.

A.2.B Details concerning the manufacturer of the investigational device Manufacturer MediTuner AB Address Peter Myndes Backe 8 118 46 Stockholm Sweden SRN SE-MF-000028534 PRRC Karlijn van Herpen Email Karlijn@asthmatuner.com Phone +46 72 853 80 46

AsthmaTuner - version number 5.4.13.5 is a CE-marked MDR, class 2b device. SpiroBank Smart or Smart One spirometer - Medical International Research (MIR) is CE-marked.

Airflow Training - Medical International Research (MIR) is CE-marked.

Traceability:

The serial numbers of AsthmaTuner spirometer (SpiroBank Smart/Smart One) are being used, can be traced through the backend of the AsthmaTuner system. The Airflow Trainers from MIR come in batches. Batch number 01 will be used in this clinical study.

Intended purpose of the investigational device:

The intended purpose of the investigational device is to support education, training, and assessment of inhalation technique for patients in clinical practice and in self-management to optimize response and adherence to self-treatment. However, the inhalation tool will be part of the AsthmaTuner system and will not be released as stand-alone device. Therefore, it will eventually be covered by the intended use of AsthmaTuner, which is:

The intended use of AsthmaTuner is to improve asthma control for adults and children over the age of 6. This is mainly done by providing information and treatment recommendations which are generated based on a patient's lung function, symptoms, and physician-prescribed treatment plan. Furthermore, AsthmaTuner facilitates the management of respiratory diseases by processing lung function and user-reported data and by providing information to adults and children over the age of 6. Any form of diagnosis of asthma or other respiratory diseases shall be done by a healthcare professional, so home use is only for indicative purposes

Populations and indications The populations and the indications for which the investigational device is intended is any subject above the age of 6 receiving pharmacological treatment through MDI or DPI devices, commonly for treatment of inflammatory respiratory conditions of asthma and/or COPD.

Necessary training based on risk assessment. According to the risk analysis assessment there are no risks which require necessary training or experience to use the inhalation app-module. Additionally, the device has instructions embedded into the software, which have been deemed safe and effective through usability testing.

Description of the current state of the art in clinical care Inhaled therapy with DPI or MDI is the cornerstone of asthma, COPD, and other respiratory diseases. Therefore, standard educational program should contain training about correct inhalation technique. The recommendations about choice and effective use of inhaler devices for educational program are presented in Table 1 according to Global Initiative for Asthma (GINA).

Table 1: Recommendations of effective use of inhaler devices according to GINA - Global Initiative for Asthma guidelines.

CHOOSE:

* Choose the most appropriate inhaler device for the patient before prescribing treatment. Consider the preferred medication, available devices, patient skills, environmental impact and costs.
* Ensure that patient have no physical or functional barriers that limit use of the inhaler.
* Avoid use of multiple different inhalers types where possible, to avoid confusion.

CHECK:

* Check inhaler technique at every opportunity
* Ask the patient to show how they use their inhaler (don't ask if they know how to use it)
* Identify any errors using device specific checklist (Table 2).

CORRECT:

* Show the patient how to use the inhaler correctly with a physical demonstrating, e.g. by using a placebo inhaler.
* Check technique again, paying attention to critical steps putting patient at risk not receiving inhaled medication. You may need to repeat this process 2-3 times within the same session for the patient to master the correct techniques [21].
* Identify any errors using a device-specific checklist (Table 2).
* Consider an alternative device only if patient cannot use the inhaler correctly after several training attempts.
* Re-check inhaler technique frequently. After initial training, errors often recur within 4-6 weeks [22].

CONFIRM:

* Clinicians should be able to demonstrate correct technique for each of the inhalers they prescribe.
* Pharmacists and nurses can provide highly effective inhaler skills training

If the patient can't use the available device(s) correctly proper education, this could be related to factors of physical dexterity, coordination, inspiratory flow and cognitive status. Different inhaler types require different inhalation techniques, so it is preferable to avoid prescribing different types of inhalers for the same patient. Furthermore, incorrect inhaler technique increases risk of severe exacerbation of asthma or COPD. Additionally, Inspiratory flow rates can be assessed with the mechanical devices. These hand-held manual meters enables assessment of PIF, in some cases through adjustable resistance selected for a relevant inhalator (DPI or MDI).

An educational and training device embedded in a patient smartphone app, shared with healthcare providers, offers novel and potentially cost-effective opportunities for healthcare providers to easily assess and monitor the performance of patients' inhalation techniques.

Justification for the design of the clinical investigation:

The choice of inhalation device is crucial for the treatment of respiratory conditions or diseases like asthma and COPD. Poor inhalation technique is a prevalent problem that makes treatment and management more difficult and costly.

The inspiratory flow is dependent on patient's technical skills and respiratory condition, as well as the resistance of the inhaler. The use of MDI or DPI requires different inhalation techniques and flows, which makes correct inhalation technique more challenging if patient use different types of inhaler devices. Healthcare providers may assess inhalation technique by observation and in addition PIF may be measured by manual meter. However, this does not capture all relevant information about patient's ability to correctly inhale medication and handle prescribed inhaler(s) and do not give instant and automated feedback on the inhalation technique to user. For instance, DPI users should reached a sufficiently high PIF within the first 0.4 seconds and MDI users inhalation time should exceed 4 seconds in adults (2-3 seconds in children) in order to optimize lung deposition of the aerosol during a low PIF. The app-based inhalation medical device gives automated feedback on inspiratory flows that are specific DPI and MDI devices. Characterization inhalation flows may also support the personalized prescription of specific inhaler for a patient. That could have significant effect on treatment response and reduction of symptoms, healthcare utilization and costs that are associated with difficulty treated asthma or COPD.

The first prototype of the inhalation app-module was tested in a clinical pilot study assessed inhalation technique in 40 schoolchildren at Astrid Lindgren Children 's Hospital, Sweden. In the study population reported 27 (71%) of 40 that their inhalation technique was improved by visualizing the inspiratory flow curve during while measuring critical endpoints of PIF, time to PIF and inhalation time in relation to selected inhaler. The respiratory nurses involved in the pilot study also reported that the automated feedback on training inhalation technique was a valuable support for education of inhalation technique in schoolchildren with asthma. The study has provided valuable information about feasibility that will be used for CE-marking the device. Therefore, we now plan for the next step to collect further information about the clinical effect on inhalation technique and the feasibility of using the device remotely in prospectively designed RCT including a larger study population with asthma and/or COPD. Integrating clinical results of the inhalation training tool in real life into a clinical evaluation and development plan as per MDCG 2024-3 section 3.4 ensures a systematic approach to validating its safety, performance, and usability. This alignment not only supports regulatory compliance but also enhances the potential for successful clinical adoption and impact on patient respiratory outcomes.

Content and relevant user interfaces of investigational device have been developed according to usability engineering to medical devices, IEC 62366-1:2015. The inventors Björn Nordlund and Henrik Ljungberg who have been involved in the design of investigational device and have also developed the AsthmaTuner, as well as founded the company MediTuner AB, which owns AsthmaTuner, through innovation programs. They are clinical health care providers themselves, working with asthma patients on a daily basis as nurse and physician at Astrid Lindgren Children's Hospital, Karolinska University Hospital in Stockholm, Sweden.

Objectives and hypotheses of the clinical investigation Our hypothesis is that the app-based investigational medical device consisting is superior for education and training of inhalation techniques in patients with asthma and COPD compared with standard care. The pre-clinical evaluation indicated the use of the investigational device is a feasible and safe for patients using inhaler(s) for treatment. The study assumption is that the investigational medical device will improve the relative rate of successful inhalation technique with at least 25% compared with control group.

Primary aim: To investigate if app-based education and training of inhalation technique improves the rate of successful inhalation techniques compared with control group at 6-12 weeks follow-up visit.

Secondary aims: To evaluate the usability and safety of the investigational device during the study period.

The claim that this clinical data can substantiate is: the inhalation app-module in AsthmaTuner is superior for education and training of inhalation techniques in patients with asthma and COPD, when compared to standard care.

There are no identified risks or anticipated adverse events that will be studied in this clinical investigation.

Design of the clinical investigation:

This confirmatory multicentre two-armed stratified randomised controlled blinded study analysing the effect of app-based education and training of inhalation technique compared with control group on subjective critical and objective endpoints of inhalation technique at 6-12 weeks follow-up visit. The study approach is intention to treat, including 80 subjects with daily therapy of DPI and/or MDI for asthma and/or COPD.

Subjective assessment of handling and inhalation techniques, adopted from Aksu F. et al. [8]. If all criteria are not deemed to correction per inhaler, including objective endpoints defines primary endpoint of subject with successful inhalation technique.

1. Shook inhaler (critical for Easyhaler). Shook the inhaler (critical for suspension)
2. Removed the cap of the inhaler correctly (critical). Removed the cap of the inhaler correctly (critical)
3. Actuated one dose / loaded capsule correctly (critical). Breathed out before slow inhalation
4. Inhaler kept in upright position (critical for some inhalers). Breathed out and away from the mouthpiece of the inhaler
5. Breathed out and away from the mouthpiece of the inhaler. Placed the inhaler mouthpiece correctly in mouth
6. Inhaler correctly placed in mouth. Inhaled with lips sealed around the mouthpiece (critical) Inhalation slow before or immediately when dose fired (critical)
7. Inhaled forcefully through the mouth after firing dose (critical) Inhaled through the mouth after dose fired (critical)
8. Inhaled without interruption (critical). Inhaler was correctly placed in mouth during the entire inhalation (critical)
9. Breath-holding more than 5 seconds after inhalation. Inhaled without interruption (critical)
10. Breathed out and away from the mouthpiece of the inhaler. Breath-holding more than 5 seconds after inhalation
11. For Handyhaler or similar, check powder drug rests in capsule, if necessary, inhale again Breathed out and away from the mouthpiece of the inhaler

Each subject in both intervention and control arm will receive standard assessment and instruction on inhalation technique. The study endpoints will be collected at the follow-up visit (6-12 weeks).

Subjects:

Inclusion criteria Subjects, age >16 years, willing to voluntarily participate in the study and give electronic written informed consent through BankID or similar service, with daily inhalation therapy through DPI and/or MDI for doctor's diagnosed asthma or COPD.

Exclusion criteria Age <16 years, no access to use BankID nor use of smartphone of type Android or iPhone, plan to stop use treatment with DPI and/or MDI the following 6-12 weeks. Medical condition affecting the ability to independently inhale or use DPI or MDI device(s).

Lost to follow-up Subjects lost to follow-up will not be replaced but the decision will be documented in the medical record. Subjects who not attend the follow-up visit 12 weeks after the baseline visit will be categorised as lost to follow-up. They will be asked through email, phone or letter to send in the medical device to the study centre with envelope they received when they received the device at baseline visit. Study sites will be informed about which subjects were lost to follow-up.

Point of enrolment and randomisation At least 80 subjects will be invited to participate in the investigation, through phone, digital meeting (Teams or Zoom or similar) or at physical at the baseline visit. The study personnel at investigational site will contact the study centre through phone to receive the randomisation assignment and study ID. The anticipated distribution is a minimum of 10 subjects per each participating investigational site.

Statistical considerations:

The analytical approach of this RCT is intention-to-treat. Additionally, a per-protocol analysis will be conducted on subjects who performed an inhalation test on average more than once per week during the study period, to evaluate the efficacy of education and training on inhalation technique between the intervention and control groups.

Primary analysis: The success rate of subjects with correct inhalation technique according to objective and subjective critical endpoints at the 6-12 weeks follow-up visit. The effect of the medical device on rate of successful inhalation technique will be determined across randomisation groups with logistic regression analysis as risk ratio (RR) with 95% confidence interval. No interim analysis will be performed.

Secondary analyses: The analysis of feasibility and the experienced benefit of inhlation education and training support will be estimated on a Likert scale from 1 (not at all) to 5 (strongly agree), and summarized as mean and median scores. Quality content analysis will assemble collected information from questionnaire and interviews of respiratory nurses together with comments from patients. Data will be presented as categories based on oral or written quotes.

Sensitivity analysis: Analyse the rate successful inhalation technique based on objective and all subjective (not only critical) endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, age >16 years, willing to voluntarily participate in the study and give electronic written informed consent through BankID or similar service, with daily inhalation therapy through DPI and/or MDI for doctor's diagnosed asthma or COPD.

Exclusion Criteria:

* Age <16 years, no access to use BankID nor use of smartphone of type Android or iPhone, plan to stop use treatment with DPI and/or MDI the following 6-12 weeks. Medical condition affecting the ability to independently inhale or use DPI or MDI device(s).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is number of subjects presenting successful inhalation techniques. | 6-12-week follow-up visit
  Defined by objective endpoints divided by:
  * DPI: PIF > 30 L/Min, time to PIF <0.5 seconds measured with the investigational device.
  * MDI: inspiration time (> 3 seconds) and PIF less than 60 L/Min measured with the investigational device.
  * Together with subjective critical endpoints, assessed by study personnel.

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Healthcare centre, Styrsö, Västra Götaland County
  - Uppsala University Hospital, Lung and Allergy Department, Uppsala
  - Healthcare Centre, Boxholm, Östergötland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armour CL, Reddel HK, LeMay KS, Saini B, Smith LD, Bosnic-Anticevich SZ, Song YJ, Alles MC, Burton DL, Emmerton L, Stewart K, Krass I. Feasibility and effectiveness of an evidence-based asthma service in Australian community pharmacies: a pragmatic cluster randomized trial. J Asthma. 2013 Apr;50(3):302-9. doi: 10.3109/02770903.2012.754463. Epub 2012 Dec 28. PMID 23270495
- [Background] Lewis A, Torvinen S, Dekhuijzen PN, Chrystyn H, Watson AT, Blackney M, Plich A. The economic burden of asthma and chronic obstructive pulmonary disease and the impact of poor inhalation technique with commonly prescribed dry powder inhalers in three European countries. BMC Health Serv Res. 2016 Jul 12;16:251. doi: 10.1186/s12913-016-1482-7. PMID 27406133
- [Background] Capstick TG, Clifton IJ. Inhaler technique and training in people with chronic obstructive pulmonary disease and asthma. Expert Rev Respir Med. 2012 Feb;6(1):91-101; quiz 102-3. doi: 10.1586/ers.11.89. PMID 22283582
- [Background] Broeders ME, Vincken W, Corbetta L; ADMIT Working Group. The ADMIT series--Issues in Inhalation Therapy. 7. Ways to improve pharmacological management of COPD: the importance of inhaler choice and inhalation technique. Prim Care Respir J. 2011 Sep;20(3):338-43. doi: 10.4104/pcrj.2011.00062. PMID 21808941
- [Background] Crompton GK, Barnes PJ, Broeders M, Corrigan C, Corbetta L, Dekhuijzen R, Dubus JC, Magnan A, Massone F, Sanchis J, Viejo JL, Voshaar T; Aerosol Drug Management Improvement Team. The need to improve inhalation technique in Europe: a report from the Aerosol Drug Management Improvement Team. Respir Med. 2006 Sep;100(9):1479-94. doi: 10.1016/j.rmed.2006.01.008. Epub 2006 Feb 21. PMID 16495040
- [Background] Basheti IA, Reddel HK, Armour CL, Bosnic-Anticevich SZ. Improved asthma outcomes with a simple inhaler technique intervention by community pharmacists. J Allergy Clin Immunol. 2007 Jun;119(6):1537-8. doi: 10.1016/j.jaci.2007.02.037. Epub 2007 Apr 16. No abstract available. PMID 17433831
- [Background] Ljungberg H, Carleborg A, Gerber H, Ofverstrom C, Wolodarski J, Menshi F, Engdahl M, Eduards M, Nordlund B. Clinical effect on uncontrolled asthma using a novel digital automated self-management solution: a physician-blinded randomised controlled crossover trial. Eur Respir J. 2019 Nov 14;54(5):1900983. doi: 10.1183/13993003.00983-2019. Print 2019 Nov. PMID 31481605
- [Background] Janssens W, VandenBrande P, Hardeman E, De Langhe E, Philps T, Troosters T, Decramer M. Inspiratory flow rates at different levels of resistance in elderly COPD patients. Eur Respir J. 2008 Jan;31(1):78-83. doi: 10.1183/09031936.00024807. Epub 2007 Sep 26. PMID 17898020
- [Background] Broeders ME, Molema J, Hop WC, Vermue NA, Folgering HT. The course of inhalation profiles during an exacerbation of obstructive lung disease. Respir Med. 2004 Dec;98(12):1173-9. doi: 10.1016/j.rmed.2004.04.010. PMID 15588037
- [Background] Richter K. Successful use of DPI systems in asthmatic patients--key parameters. Respir Med. 2004 Oct;98 Suppl B:S22-7. doi: 10.1016/j.rmed.2004.07.013. PMID 15481285
- [Background] Bronsky EA, Grossman J, Henis MJ, Gallo PP, Yegen U, Della Cioppa G, Kottakis J, Mehra S. Inspiratory flow rates and volumes with the Aerolizer dry powder inhaler in asthmatic children and adults. Curr Med Res Opin. 2004;20(2):131-7. doi: 10.1185/030079903125002793. PMID 15006006
- [Background] Boulet LP, FitzGerald JM, Levy ML, Cruz AA, Pedersen S, Haahtela T, Bateman ED. A guide to the translation of the Global Initiative for Asthma (GINA) strategy into improved care. Eur Respir J. 2012 May;39(5):1220-9. doi: 10.1183/09031936.00184511. Epub 2012 Jan 26. PMID 22282546
- [Background] Aksu F, Sahin AD, Sengezer T, Aksu K. Effect of training by a physician on dynamics of the use of inhaler devices to improve technique in patients with obstructive lung diseases. Allergy Asthma Proc. 2016 Sep;37(5):98-102. doi: 10.2500/aap.2016.37.3969. Epub 2016 May 9. PMID 27164509
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary. Eur Respir J. 2017 Mar 6;49(3):1700214. doi: 10.1183/13993003.00214-2017. Print 2017 Mar. PMID 28182564
- [Background] Jansson SA, Ronmark E, Forsberg B, Lofgren C, Lindberg A, Lundback B. The economic consequences of asthma among adults in Sweden. Respir Med. 2007 Nov;101(11):2263-70. doi: 10.1016/j.rmed.2007.06.029. Epub 2007 Aug 6. PMID 17689234

DOCUMENTS (1):
  • Study Protocol (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT07145632/Prot_000.pdf